CLINICAL TRIAL: NCT06062862
Title: Effect of Breather on Hospital Stay in Patients With Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Mousa Galeb, Lecturer at the Department of Physical Therapy for Cardiovascular /Respiratory Disorders and Geriatrics Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hospital Acquired pneumonia
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pneumonia Hospital Acquired
Keywords: Incentive spirometry,Breather, Acquired pneumonia, Arterial blood gases
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Intervention Model Description: Group A (study group): 30 patients (15 males and 15 females) will receive respiratory training using incentive spirometer in addition to traditional chest physiotherapy, 3 sessions per day, for 2 weeks.
  Group B (study goup): 30 patients (15 males and 15 females) will receive respiratory training using the breather in addition to traditional chest physiotherapy, 3 sessions per day, for 2 weeks.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Incentive Spirometer group (Active Comparator): The respiratory muscle training program has the following parameters: Duration: 20 minutes per session, Intensity: Clinical adjustment of training intensity based on actual participants' status across session time, holding time, and repetitions. Frequency: 30 per set, with each is 5-6 times. The procedure for the respiratory muscle training program is as follows: a deep slow inspiration while lips fitted around mouthpiece. Visual feedback is provided to the patient, such as a ball rising to a preset marker, to motivate them during the exercise. The patient is instructed to get the planned flow at preset amount. The patient is asked to maintain breathing in along 2-3 seconds. These guidelines should be followed during respiratory muscle training
  Interventions: Device: The Incentive Spirometer
- The Breather Respiratory Muscle Trainer group (Active Comparator): Utilizing a pre-session checklist can improve the success rate of using the breather for respiratory muscle training. The following items should be included in the checklist: Check the patient's posture, ensuring that they are in a comfortable crook lying or sitting position, initial easiest resistances by manipulating both dials to one, ensure the patient is using the diaphragmatic breathing technique, as this is crucial for the proper use of the breather, and make sure that the patient secures lips on mouthpiece.
  Interventions: Device: The breather respiratory muscle training device

INTERVENTIONS:
Device: The Incentive Spirometer — Tri-flow device flow-oriented incentive spirometer .
  Arms: The Incentive Spirometer group
Device: The breather respiratory muscle training device — The breather respiratory muscle training device which allows for adjustable levels of resistance using easy-to-read dials, which allows to adjust the device to the settings require
  Arms: The Breather Respiratory Muscle Trainer group

SUMMARY:
Acquired pneumonia is a sever medical condition that addressed as life-threatening issue require intensive care. Medical Breather device permits activating and strengthening of both inspiratory and expiratory musculatures; thus, it could be useful for pneumatic patients. The aim of the study is to investigate breather effect on hospital stay in pneumatic patients.

DETAILED DESCRIPTION:
Sixty participants diagnosed with acquired pneumonia '30 women, 30 men; selected from chest department of Kasr Alaini Intensive Care Unit (ICU) at Cairo University. They were randomly allocated into equal groups; Group A received respiratory training via incentive spirometer, and traditional chest physiotherapy; and Group B received respiratory training via Breather, and traditional chest physiotherapy. both received 3 session daily/2 weeks. Diaphragmatic excursion, Respiratory Distress Observation Scale, and ICU discharge were assessed pre and post treatment.

Careful recruitment of participants based on the study criteria by both ICU resident and PT consultant. Identified inclusive criteria include conscious both genders aged 30- 40 years old with BMI ranged from 25 to5 29.9 Kg/m2 had an acquired pneumonia with a mild hypoxemia (O2 saturation was 90 - 95%). Aware participants whom cooperated through accurate understand and perform instructions. Excluding patients through identified inclusive criteria that if they had a history of any malignant tumors, hearing impairment or mental disorder, auto-immune diseases, a history of any surgical transplantation, unstable hemodynamics, rib fracture, a history of neuromuscular disease, spinal injuries, or BMI > 30 Kg/m2. Also, patients receiving mechanical ventilation, or whom require MV, but contraindicated for rehabilitation i.e., pulmonary emboli were excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty patients of both sexes from intensive care unit, Cairo University Hospitals.
2. Their age ranged from 30 to 40 years old.
3. Their BMI were from 25 - 29.9 Kg/m2.
4. Their oxygen saturation 90 - 95% (mild hypoxemia) conscious level.

Exclusion Criteria:

1. Patient with a history of any malignant tumors. 2. Patients with hearing impairment or mental disorder. 3. Patients with auto-immune diseases. 4. Patients with a history of any surgical transplantation. 5. Patients with hemo-dynamically unstable patients. 6. Patients with rib fracture. 7. Patients with history of neuromuscular disease. 8. Patients with spinal injuries. 9. Patients with BMI > 30 Kg/m2. 10. Patients receiving mechanical ventilation.

-

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
arterial blood gases (ABG) | Pre and post treatment after 2 weeks
  * potential of hydrogen( pH )(7.35-7.45).
  * the partial pressure of carbon dioxide in arterial blood.(PaCO2 )(35-45 mmHg).
  * Bicarbonate (HCO3)(22-28 meq/L).
  * arterial oxygen saturation (SaO2) (95-100%).
  * pH (7.35-7.45).
  * PaCO2 (35-45 mmHg).
  * HCO3 (22-28 meq/L).
  * SaO2 (95-100%). . Sample was taken from the radial artery to measure the following parameters6: 7.35-7.45 PH, 35-45 mmHg PaCO2, 22-28 meq/L HCO3, and 95-100% SaO2.
Diaphragmatic excursion | Pre and post treatment after 2 weeks
  measured diaphragmatic movement for each subject by using the Diaphragmatic ultrasound at 3.5-5MHz probe that aimed at midclavicular line under rib cage aiming posterior 3rd of hemi diaphragm.
Respiratory distress observation scale (RDOS) | Pre and post treatment after 2 weeks
  evaluate severity and discomfort experienced by patients who are unable to communicate their dyspnea levels during monitoring for palliative sedation therapy .
  RDOS score of less than 3 indicates that the patient is breathing comfortably, d) an RDOS value ≥3 means respiratory distress that require palliative measures, and e) higher RDOS scores indicate a worsening of the patient's condition.
The National Early Warning Score 2 (NEWS2) | Pre and post treatment after 2 weeks
  ) scoring system for evaluating hospital discharge. It measures six physiological items; respiration and pulse rates, O2 saturation, systolic blood pressure, consciousness level or recent onset confusion, also temperature 9. Each parameter is allocated a score of 0, 1, 2, or 3, elevated values indicate that is far away from normal values.
  1. Low risk (aggregate score of 1-4).
  2. Low to moderate '3 in a single item' risk.
  3. Moderate risk (aggregate score of 5-6).
  4. Maximum risk (≥7 value). Critical team of care should perform an emergency assessment, often advice transfer case to a higher dependency unit, and
  5. a NEWS2 ≥ 0 i.e., no change, warrants a minimum twice daily check that be a routine monitoring.
Body mass index (BMI ) | Pre and post treatment after 2 weeks
  Ranged from 25 to 29.9 Kg/m2.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Lanks CW, Musani AI, Hsia DW. Community-acquired Pneumonia and Hospital-acquired Pneumonia. Med Clin North Am. 2019 May;103(3):487-501. doi: 10.1016/j.mcna.2018.12.008. Epub 2019 Mar 7. PMID 30955516
- [Background] Klompas M. Prevention of Intensive Care Unit-Acquired Pneumonia. Semin Respir Crit Care Med. 2019 Aug;40(4):548-557. doi: 10.1055/s-0039-1695783. Epub 2019 Oct 4. PMID 31585480